CLINICAL TRIAL: NCT05236608
Title: A Phase 1b/2 Study to Evaluate the Combination of Nivolumab (Anti PD1 Monoclonal Ab) With ADG106 (4-1-BB Agonist Monoclonal Ab) in Metastatic NSCLC After Progression With antiPD1 Therapy and Platinum-based Chemotherapy (ADIVO Lung Study)
Brief Title: A Study to Evaluate the Combination of Nivolumab With ADG106 in Metastatic NSCLC
Acronym: ADIVO Lung
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Adagene Inc (Industry); Bristol-Myers Squibb (Industry); Singapore Translational Cancer Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STCC-02; CA209-63C (Other: BMS); ADG106-T6001 (Other: Adagene)
Record Dates: First submitted 2021-10-11; First posted 2022-02-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab and ADG106 (Experimental): Eligible patients will receive nivolumab and ADG106 by IV infusion according to the study phases below.
  Phase 1b:
  3 evaluable patients will be treated at the starting dose, and assessed for tolerability over the first cycle. Treatment related dose-limiting toxicities (DLT) will determine the next dose level to be studied. Dose escalation will follow the 3 + 3 study dose titration design.
  Phase 2:
  The dose of ADG106 given together with nivolumab will be the recommended dose in combination with nivolumab determined in phase 1b.
  Interventions: Drug: Nivolumab; Drug: ADG106

INTERVENTIONS:
Drug: Nivolumab — Administered together with ADG106 via intravenous infusion.
  Other Names: Opdivo
Drug: ADG106 — Administered as an intravenous infusion over 90 minutes.

SUMMARY:
This is an open label, non-randomised phase 1b/2 study including patients with non-small cell lung cancer who have progressed after treatment with immune checkpoint inhibitors (anti PD1/PDL1 with or without CTLA4 inhibitors) and platinum-based chemotherapy. The study medications include nivolumab, an anti-PD1 inhibitor and ADG106, an agonist antibody of 4-1-BB.

The investigators hypothesize that the combination of nivolumab and ADG106 would be tolerable, and demonstrate significant clinical anti-tumour activity in patients with NSCLC that has failed antiPD1/antiPDL1 immunotherapy and standard platinum-based chemotherapy. The investigators propose to conduct a phase 1b/2 study to investigate this strategy.

ELIGIBILITY:
Inclusion Criteria:

1. For Phase 1b: Patients with histologically or cytologically confirmed solid malignancies

   1. who are refractory to standard of care treatment OR
   2. have no standard of care treatment of curative potential.

   For Phase 2: Patients with histologically or cytologically confirmed stage 4 or recurrent NSCLC (per IASLC classification) who have progression of disease
   1. after treatment with antiPD1/PDL1 with CTLA4 inhibitors and at least one platinum-based chemotherapy OR
   2. after treatment with antiPD1/PDL1 without CTLA4 inhibitors and at least one platinum-based chemotherapy
2. The participant (or legally acceptable representative if applicable) provides written consent for the trial.
3. Participants who are at least 21 years of age on the day of signing informed consent.
4. Eastern Cooperative Group (ECOG) Performance Status 0-1
5. Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Previously irradiated lesions is considered measurable if they show progression after completion of radiation therapy.
6. Have adequate organ function. Specimens must be collected within 7 days prior to the start of study treatment.
7. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential OR
   2. A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study medication.
8. A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
9. Willing to participate in the translational blood and tissue collection studies.
10. Availability of archival formalin-fixed, paraffin-embedded (FFPE) tumour tissue block or unstained tumour tissue specimens if fresh tumour biopsy is not feasible.

Exclusion Criteria:

1. Has received prior systemic anti-cancer therapy including investigational agents within 3 weeks prior to enrolment.

   Note: Participants must have recovered from all AEs to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
2. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
3. Prior severe immune adverse events of grade 3 or 4 to antiPD1/PDL1 therapy. These include interstitial pneumonitis.
4. Has a known history of active TB (Mycobacterium tuberculosis).
5. Known allergy to any of the ingredients of ADG106 (succinic acid, arginine, polysorbate 80 and hydrochloric acid) in the formulation or known allergy to any related class of compounds (note: polysorbate 80 is an ingredient in docetaxel).
6. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast or cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.
8. Known brain metastases or leptomeningeal metastases that are not adequately treated and require corticosteroids of > 10mg daily prednisolone or its equivalent at least 7 days prior to study treatment start date.
9. Has an active infection requiring systemic therapy.
10. History of having received a live virus vaccination (eg yellow fever, MMR, nasal flu, chicken pox or Zostavax) in the past 1 month.
11. Subjects with underlying hemoglobinopathies (e.g., thalassemia).
12. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
13. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrolment. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
14. Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Subjects with active hepatitis B (positive hepatitis B surface antigen [HBsAg] with detectable serum HBV DNA) or HCV (hepatitis C virus) [positive HCV RNA]). Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to enrolment. HBsAg positive carriers or those patients with undetectable serum HBV DNA and on antiviral therapy are eligible to participate. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
17. Known history of testing positive for human immunodeficiency virus (HIV) or Known history of testing positive for known acquired immunodeficiency syndrome (AIDS). NOTE: Testing for HIV must be performed at sites where mandated locally.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 45 months
  Adverse events profile, safety profile of the combination of ADG106 and nivolumab according to the NCI Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Objective response rate | 24 months
  Objective response rate (CR + PR) using RECIST 1.1 of the combination of ADG106 and nivolumab in patients with metastatic NSCLC that have progressed after antiPD1/PDL1 treatment and platinum-based chemotherapy (phase 2).

SECONDARY OUTCOMES:
Progression free survival at 6 months | 6 months
  Progression free survival at 6 months of the combination of ADG106 and nivolumab in patients with metastatic NSCLC that have progressed after antiPD1/PDL1 treatment and platinum-based chemotherapy (phase 2) and the irRECIST objective response rate.
Area Under the Curve [AUC] | Baseline until Cycle 2 Day 1, each cycle is 21 days
  Pharmacokinetics of nivolumab/ADG106 will be measured using blood samples collected at specify timepoint
Maximum Plasma Concentration [Cmax] | Baseline until Cycle 2 Day 1, each cycle is 21 days
  Pharmacokinetics of nivolumab/ADG106 will be measured using blood samples collected at specify timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez-Paulete AR, Labiano S, Rodriguez-Ruiz ME, Azpilikueta A, Etxeberria I, Bolanos E, Lang V, Rodriguez M, Aznar MA, Jure-Kunkel M, Melero I. Deciphering CD137 (4-1BB) signaling in T-cell costimulation for translation into successful cancer immunotherapy. Eur J Immunol. 2016 Mar;46(3):513-22. doi: 10.1002/eji.201445388. Epub 2016 Feb 9. PMID 26773716
- [Result] Costantini A, Corny J, Fallet V, Renet S, Friard S, Chouaid C, Duchemann B, Giroux-Leprieur E, Taillade L, Doucet L, Nguenang M, Jouveshomme S, Wislez M, Tredaniel J, Cadranel J. Efficacy of next treatment received after nivolumab progression in patients with advanced nonsmall cell lung cancer. ERJ Open Res. 2018 Apr 20;4(2):00120-2017. doi: 10.1183/23120541.00120-2017. eCollection 2018 Apr. PMID 29692997
- [Result] Freeman AT, Lesperance M, Wai ES, Croteau NS, Fiorino L, Geller G, Brooks EG, Poonja Z, Fenton D, Irons S, Ksienski D. Treatment of non-small-cell lung cancer after progression on nivolumab or pembrolizumab. Curr Oncol. 2020 Apr;27(2):76-82. doi: 10.3747/co.27.5495. Epub 2020 May 1. PMID 32489249
- [Result] Qi X, Li F, Wu Y, Cheng C, Han P, Wang J, Yang X. Optimization of 4-1BB antibody for cancer immunotherapy by balancing agonistic strength with FcgammaR affinity. Nat Commun. 2019 May 20;10(1):2141. doi: 10.1038/s41467-019-10088-1. PMID 31105267